CLINICAL TRIAL: NCT02670382
Title: Role of EPA and DHA in Fish Oil on Inflammation and Lipoprotein Metabolism
Brief Title: Role of Eicosapentaenoic Acid (EPA) and Docosahexaenoic Acid (DHA) on Inflammation and Lipids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Stefania lamon-Fava, Scientist I, Associate Professor, Tufts University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2845
Record Dates: First submitted 2015-12-23; First posted 2016-02-01 (Estimated); Results first posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Eicosapentaenoic Acid; Sunflower Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- EPA intervention (Experimental): Subjects randomized to receive 3000 mg EPA/day, provided as EPA 750 mg/capsule will be instructed to take 2 capsules by mouth in the morning and 2 in the evening with meals for 10 weeks.
  Interventions: Dietary Supplement: EPA
- DHA intervention (Experimental): Subjects randomized to 3000 mg DHA/day provided as DHA 750 mg/capsule will instructed to take 2 capsules by mouth in the morning and 2 in the evening with meals for 10 weeks.
  Interventions: Dietary Supplement: DHA
- Placebo (Placebo Comparator): 3000 mg high oleic acid sunflower oil/day; 750 mg high oleic acid sunflower oil/capsule; subjects instructed to take 2 capsules by mouth in the morning and 2 in the evening with meals during 4 week long lead-in phase.
  Interventions: Dietary Supplement: sunflower oil

INTERVENTIONS:
Dietary Supplement: EPA — 10 week supplementation
  Other Names: eicosapentaenoic acid
  Arms: EPA intervention
Dietary Supplement: DHA — 10 week supplementation
  Arms: DHA intervention
Dietary Supplement: sunflower oil — 4-week lead-in
  Arms: Placebo

SUMMARY:
The objective of this study is to provide critical information regarding both common and distinctive roles of EPA and DHA in systemic inflammation and lipid metabolism.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind, crossover study of the effects of EPA and DHA on inflammation and lipid metabolism in 24 men and women with metabolic syndrome. The study will characterize the effects of EPA alone and DHA alone, relative to each other and to placebo, on plasma biomarkers of inflammation, inflammatory cell activation and gene expression, and plasma lipid and lipoprotein levels.

ELIGIBILITY:
Inclusion criteria:

* fasting plasma TG levels between 150 and 500 mg/dL
* C-reactive protein (CRP) levels ≥2 µg/mL
* at least one of the following criteria for the definition of metabolic syndrome:

  * abdominal obesity (waist circumference >40 inches in men and >35 inches in women),
  * hypertension (blood pressure ≥130/≥85 mmHg or use of anti-hypertensive medications), and
  * fasting glucose ≥110 mg/dL.

Exclusion criteria:

* high-fish diets (>2 fish meals/week)
* taking fish oil supplements or supplements containing EPA or DHA
* allergy to sardines
* allergy to sunflower oil
* regular use of anti-inflammatory medications (NSAID, COX inhibitors, corticosteroids)
* anticoagulant therapy
* alcohol consumption >7 drinks/week
* uncontrolled thyroid dysfunction
* insulin-dependent type 2 diabetes mellitus
* kidney or liver disease
* smoking
* alterations in coagulation
* use of lipid altering medications

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2020-05 (Actual); Study Completion 2020-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefania Lamon-Fava, PhD, Principal Investigator — Tufts University
Locations (1):
- Jean Mayer Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
The objective of this study is to provide critical information regarding both common and distinctive roles of the omega-3 fatty acids EPA and DHA in systemic inflammation and lipid metabolism.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 405 subjects were screened for eligibility at the Metabolic Research Unit of the Human Nutrition Research Center on Aging at Tufts Unoversity
Pre-assignment Details: 24 subjects met the inclusion criteria and were enrolled into the study. 3 subjects dropped off during the placebo lead-in phase of the study
Groups:
- Placebo, Then EPA, Then DHA: 3000 mg high oleic acid sunflower oil/day during 4-week lead-in phase; then participants received 3000 mg pure EPA for 10 weeks; then washout of 10 weeks; then pure DHA 3000 mg/day Placebo and EPA and DHA capsules provided as 750 mg/capsule; subjects instructed to take 2 capsules by mouth in the morning and 2 in the evening
- Placebo, Then DHA, and Then EPA: 3000 mg high oleic acid sunflower oil/day during 4-week lead-in phase; then participants received 3000 mg pure DHA for 10 weeks; then washout of 10 weeks; then pure EPA 3000 mg/day Placebo and DHA and EPA capsules provided as 750 mg/capsule; subjects instructed to take 2 capsules by mouth in the morning and 2 in the evening
Period: Placebo lead-in Phase
Arm/Group | Placebo, Then EPA, Then DHA | Placebo, Then DHA, and Then EPA
Started | 12 | 12
Completed | 10 (Two enrolled subjects randomized to receive EPA as the first intervention decided to stop participation during the placebo lead-in phase. Therefore, only 10 subjects continued to the EPA and then DHA supplementation phases. No data were collected from these two subjects.) | 11 (One enrolled subjects randomized to receive EDHA as the first intervention decided to stop participation during the placebo lead-in phase. Therefore, only 11 subjects continued to the DHA and then EPA supplementation phases. No data were collected from this subject.)
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1
Period: First Active Intervention
Arm/Group | Placebo, Then EPA, Then DHA | Placebo, Then DHA, and Then EPA
Started | 10 (Only 10 of the 12 enrolled subjects randomized to receive EPA as the first supplementation completed the lead-in placebo phase and then entered the EPA supplementation phase.) | 11 (Only 11 of the 12 enrolled subjects randomized to receive DHA as the first supplementation completed the lead-in placebo phase and then entered the EDHA supplementation phase.)
Completed | 10 | 11
Not Completed | 0 | 0
Period: Second Active Intervention
Arm/Group | Placebo, Then EPA, Then DHA | Placebo, Then DHA, and Then EPA
Started | 10 | 11
Completed | 10 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Baseline characteristic, defined as end of lead-in phase
Arm/Group | All Participants
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] — years, continuous variable
  years | 62 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 32.20 (6.61)
C reactive protein [Mean (Standard Deviation); unit: microg/mL] | 6.0 (3.4)
Glucose [Mean (Standard Deviation); unit: mg/dL] | 99 (11)
triglycerides [Mean (Standard Deviation); unit: mg/dL] | 145 (51)

OUTCOME MEASURES:

1. Primary Outcome: Interleukin-6 (IL-6)
Description: plasma levels in pg/mL
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | EPA Intervention | DHA Intervention
Number analyzed (Participants) | 21 | 21 | 21
pg/mL | 0.96 (0.56) | 1.01 (0.51) | 0.99 (0.77)
Statistical Analysis 1: Comparison: Placebo vs EPA Intervention; Test type: Superiority; p = 0.33, Mixed Models Analysis; mean values, log transformed
Statistical Analysis 2: Comparison: Placebo vs DHA Intervention; Test type: Superiority; p = 0.92, Mixed Models Analysis; mean difference, log transformed values
Statistical Analysis 3: Comparison: EPA Intervention vs DHA Intervention; Test type: Superiority; p = 0.44, Mixed Models Analysis; mean difference, log transformed values

2. Primary Outcome: Tumor Necrosis Factor Alpha (TNF-alpha)
Description: plasma levels in pg/mL
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | EPA Intervention | DHA Intervention
Number analyzed (Participants) | 21 | 21 | 21
pg/mL | 2.38 (0.54) | 2.48 (0.64) | 2.47 (0.76)
Statistical Analysis 1: Comparison: Placebo vs EPA Intervention; Test type: Superiority; p = 0.34, Mixed Models Analysis; mean difference, log transformed values
Statistical Analysis 2: Comparison: Placebo vs DHA Intervention; Test type: Superiority; p = 0.50, Mixed Models Analysis; mean difference, log transformed values
Statistical Analysis 3: Comparison: EPA Intervention vs DHA Intervention; Test type: Superiority; p = 0.83, Mixed Models Analysis; mean differences, log transformed values

3. Primary Outcome: Low Density Lipoprotein Cholesterol (LDL-C)
Description: plasma levels in mg/dL
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | EPA Intervention | DHA Intervention
Number analyzed (Participants) | 21 | 21 | 21
mg/dL | 130 (26) | 136 (26) | 140 (32)
Statistical Analysis 1: Comparison: Placebo vs EPA Intervention; Test type: Equivalence — primary hypothesis is that EPA will not differ from placebo; p = 0.10, Mixed Models Analysis; mean differences
Statistical Analysis 2: Comparison: Placebo vs DHA Intervention; Test type: Superiority; p = 0.005, Mixed Models Analysis; mean difference
Statistical Analysis 3: Comparison: EPA Intervention vs DHA Intervention; Test type: Superiority; p = 0.17, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: adeverse events were collected during the participation of study subjects, equivalent to 34 weeks
Arm/Group | EPA Intervention | DHA Intervention | Placebo
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21 | 1/21
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EPA Intervention (N=21) | DHA Intervention (N=21) | Placebo (N=21)
gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) — subjects experienced left ankle swelling 4 days after starting placebo lead in phase
hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — subjects had blood pressure 177/80 at visit

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-21): https://cdn.clinicaltrials.gov/large-docs/82/NCT02670382/Prot_SAP_000.pdf